CLINICAL TRIAL: NCT00005599
Title: Phase II Trail of Bryostatin-1 and Paclitaxel in Patients With Advanced Esophageal Cancer
Brief Title: Bryostatin 1 Plus Paclitaxel in Treating Patients With Locally Advanced or Metastatic Esophageal Cancer or Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067712; MSKCC-99094; MSKCC-FDR001826; NCI-250
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2004-08

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — bryostatin 1; Paclitaxel

INTERVENTIONS:
Drug: bryostatin 1
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of bryostatin 1 and paclitaxel in treating patients who have locally advanced or metastatic esophageal cancer or stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete and partial response rates in patients with unresectable or metastatic esophageal cancer or carcinoma of the gastroesophageal junction treated with sequential paclitaxel and bryostatin 1.
* Determine the toxicity of this regimen in this patient population.
* Determine the survival of patients after treatment with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Examine pre- and post-treatment tissue biopsies for markers of apoptosis in selected patients.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 1 hour on day 1 and bryostatin 1 IV over 24 hours on day 2 weekly for 2 weeks. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

Quality of life is assessed at baseline, after courses 1 and 2, and then after every 2 courses thereafter.

PROJECTED ACCRUAL: A total of 19-33 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma or adenocarcinoma of the esophagus or carcinoma of the gastroesophageal (GE) junction

  * If tumor extends below GE junction into the proximal stomach, 50% of the tumor must involve the esophagus or GE junction
  * No gastric cancer with only a minor involvement of GE junction or distal esophagus
* Locally advanced and considered surgically unresectable or metastatic
* Measurable disease

  * Accurately measured in at least 1 dimension as at least 20 mm with conventional techniques or at least 10 mm with spiral CT scan
  * No truly nonmeasurable lesions only:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusions
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No history of active angina
* No myocardial infarction within the past 6 months
* No history of significant ventricular arrhythmia requiring medication with antiarrhythmics
* Well-controlled atrial fibrillation on standard management allowed

Pulmonary:

* DLCO at least 60%

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation
* No preexisting neurotoxicity of grade 3 or greater
* No serious concurrent infection or nonmalignant medical illness that is uncontrolled or whose control may be jeopardized by complications of study therapy
* No concurrent psychiatric disorders that would preclude study compliance
* No other active malignancy within the past 5 years except:

  * Nonmelanoma skin cancer
  * Carcinoma in situ of the cervix
  * History of T1a or b prostate cancer (detected incidentally at transurethral resection of prostate [TURP] and comprising less than 5% of resected tissue) provided prostate-specific antigen remained normal since TURP removal
* HIV negative
* No other concurrent medical condition that would preclude study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* Recovered from prior chemotherapy
* No more than 1 prior neoadjuvant or adjuvant regimen for esophageal cancer
* No prior taxanes for esophageal cancer
* No prior bryostatin 1 for esophageal cancer
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy allowed provided recent evidence of disease progression if indicator lesion is within prior radiation field
* Recovered from prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-02; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York

REFERENCES:
- [Result] Ku GY, Ilson DH, Schwartz LH, Capanu M, O'Reilly E, Shah MA, Kelsen DP, Schwartz GK. Phase II trial of sequential paclitaxel and 1 h infusion of bryostatin-1 in patients with advanced esophageal cancer. Cancer Chemother Pharmacol. 2008 Oct;62(5):875-80. doi: 10.1007/s00280-008-0677-y. Epub 2008 Feb 13. PMID 18270704